CLINICAL TRIAL: NCT03966612
Title: Study and Monitoring of Multiple Endocrine Neoplasia Type 1
Acronym: NEM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GOUDET 2018
Record Dates: First submitted 2019-01-11; First posted 2019-05-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: MEN1
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Questionnaires about:
  * Socio-professional situation
  * Lifestyle
  * Health
  * NME 1
  * specific breast cancer survey
  * Imaging

SUMMARY:
Multiple Endocrine Neoplasia Type I (MEN1) is a rare autosomal dominant disorder, predisposing sufferers to the development of endocrine tumors. The three most commont endocrine disorders of MEN1 are the secretory tumours of the parathyroid, pituitary gland and pancreas, in addition to which other tumours may be observed.

The diagnosis of MEN1 is essential for 1) appropriate therapeutic management of proven endocrine disorders, 2) screening for other endocrine and non-endocrine tumours, 3) family screening of affected relatives and 4) monitoring of patients who have been diagnosed. Undiagnosed MEN1 is one of the reasons for therapeutic failure in the management of endocrine damage. Detection is therefore of major importance, and any improvement in early diagnosis can improve management.

The natural history of the disease in all its clinical forms remains poorly understood, with published studies of selected or small populations. There are still clinical forms that are difficult to link to the syndrome. These clinical forms need to be specified in order to ensure optimal management. Only a large cohort will lead to the identification of the various forms of this condition and clarify its prognosis.

ELIGIBILITY:
Inclusion Criteria:

SYMPTOMATIC PATIENTS

* person (adult or minor) who has not opposed participation
* if the patient is a minor, the parents must not oppose their child's participation,
* at least two of the three main types of lesions (parathyroid, pancreas, pituitary gland)
* OR a known isolated tumor, main type or not, associated with the gene mutation of the NEM1 locus on chromosome 11q13
* OR an isolated tumor, main type or not, in an individual with a confirmed family history of NEM1

ASYMPTOMATIC PATIENTS WITH A MUTATION

- Presence of a characteristic mutation of NEM1

Exclusion Criteria: NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in consultation
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
risk of occurrence of each type of MEN1 related tumors | Through study completion, an average of 10 years
  risk of occurrence of each type of MEN1 related tumors in patients with confirmed MEN-1
genotype-phenotype correlation : association of specific mutations (genotype) with the clinical manifestations (phenotype) | Through study completion, an average of 10 years
overall survival | Through study completion, an average of 10 years
specific survival and life expectancy | Through study completion, an average of 10 years
age at Men1 diagnosis globally and according to the initial presentation | Through study completion, an average of 10 years
treatment description of each type of MEN1 related tumors as well as their impact on survival and on disease control | Through study completion, an average of 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France